CLINICAL TRIAL: NCT01414634
Title: Establish Tolerance in Multiple Sclerosis With Peptide-coupled, Peripheral Blood Mononuclear Cells - A MRI-controlled, Single Center, Phase I Trial in Relapsing-remitting MS Patients
Brief Title: Establish Tolerance In MS With Peptide-Coupled, Peripheral Blood Mononuclear Cells
Acronym: ETIMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: inims-oo1
Record Dates: First submitted 2011-08-08; First posted 2011-08-11 (Estimated); Results first posted 2015-04-08 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- ETIMS 1x10^3 (Experimental): The drug product consists of autologous peripheral blood mononuclear cells that have been chemically coupled with seven myelin peptides and resuspended in autologous plasma. This patient receives 1x10^3 cells.
  Interventions: Biological: ETIMS
- ETIMS 1x10^5 (Experimental): The drug product consists of autologous peripheral blood mononuclear cells that have been chemically coupled with seven myelin peptides and resuspended in autologous plasma. This patient receives 1x10^5 cells.
  Interventions: Biological: ETIMS
- ETIMS 1x10^7 (Experimental): The drug product consists of autologous peripheral blood mononuclear cells that have been chemically coupled with seven myelin peptides and resuspended in autologous plasma. This patient receives 1x10^7 cells.
  Interventions: Biological: ETIMS
- ETIMS 1x10^8 (Experimental): The drug product consists of autologous peripheral blood mononuclear cells that have been chemically coupled with seven myelin peptides and resuspended in autologous plasma. This patient receives 1x10^8 cells.
  Interventions: Biological: ETIMS
- ETIMS 5x10^8 (Experimental): The drug product consists of autologous peripheral blood mononuclear cells that have been chemically coupled with seven myelin peptides and resuspended in autologous plasma. This patient receives 5x10^8 cells.
  Interventions: Biological: ETIMS
- ETIMS 1x10^9 (Experimental): The drug product consists of autologous peripheral blood mononuclear cells that have been chemically coupled with seven myelin peptides and resuspended in autologous plasma. This patient receives 1x10^9 cells.
  Interventions: Biological: ETIMS
- ETIMS 2.5x10^9 (Experimental): The drug product consists of autologous peripheral blood mononuclear cells that have been chemically coupled with seven myelin peptides and resuspended in autologous plasma. This patient receives 2.5x10^9 cells.
  Interventions: Biological: ETIMS
- ETIMS 3x10^9 (Experimental): The drug product consists of autologous peripheral blood mononuclear cells that have been chemically coupled with seven myelin peptides and resuspended in autologous plasma. This patient receives 3x10^9 cells.
  Interventions: Biological: ETIMS

INTERVENTIONS:
Biological: ETIMS — injection of peptide-coupled PBMC by i.v. infusion

SUMMARY:
Open-label, single center, phase I clinical trial to assess the safety, tolerability and preliminary efficacy and in vivo mechanisms of action of i.v. administration of autologous peripheral blood mononuclear cell (PBMC) chemically coupled with a cocktail containing seven immunodominant myelin peptides to which T cell responses are demonstrable in early RR MS patients.

DETAILED DESCRIPTION:
Open-label, single center, phase I dose-escalation study to assess the safety, tolerability and preliminary efficacy and in vivo mechanisms of action of a single infusion of autologous peripheral blood mononuclear cells chemically coupled with seven myelin peptides (MOG1-20, MOG35-55, MBP13-32, MBP83-99, MBP111-129, MBP146-170, and PLP139-154) in Multiple Sclerosis patients who were off-treatment for standard therapies. Neurological, magnetic resonance imaging, laboratory, and immunological examinations were performed to assess the safety, tolerability, and in vivo mechanisms of action of this regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 55 years.
2. Patients with relapsing-remitting (Phase I/II) or secondary progressive MS (Phase I) according to published criteria
3. EDSS score between 1 and 5.5.
4. Patients are off-treatment for standard therapies (interferon-beta, glatiramer acetate, natalizumab, mitoxantrone)
5. Patients are able to provide written, informed consent prior to any testing under this protocol, including screening and baseline investigations that are not considered part of routine patient care.
6. Disease duration ≤ 5 years (Only Phase II)

Exclusion Criteria:

1. Diagnosis of secondary-progressive (Phase II) or primary-progressive MS, as defined by published diagnostic criteria.
2. Abnormal screening/baseline blood tests exceeding any of the limits defined
3. Pregnant or breast-feeding female.
4. History or signs of immunodeficiency.
5. Concurrent clinically significant (as determined by the investigators) cardiac, immunological, pulmonary, neurological, renal or other major disease.
6. Splenectomy
7. History of HIV or positive HIV antibody testing
8. Serology indicating active Hepatitis B or C infection.
9. Patients with cognitive impairments who are unable to provide written, informed consent prior to any testing under this protocol, including screening and baseline investigations that are not considered part of routine patient care

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Heesen, MD, Principal Investigator — Department of Neurology, University Clinic Eppendorf (UKE)

REFERENCES:
- [Result] Lutterotti A, Yousef S, Sputtek A, Sturner KH, Stellmann JP, Breiden P, Reinhardt S, Schulze C, Bester M, Heesen C, Schippling S, Miller SD, Sospedra M, Martin R. Antigen-specific tolerance by autologous myelin peptide-coupled cells: a phase 1 trial in multiple sclerosis. Sci Transl Med. 2013 Jun 5;5(188):188ra75. doi: 10.1126/scitranslmed.3006168. PMID 23740901

RESULTS

PARTICIPANT FLOW:
Groups:
- ETIMS 1x10^3; ETIMS 1x10^5; ETIMS 1x10^7; ETIMS 1x10^8; ETIMS 5x10^8; ETIMS 1x10^9; ETIMS 2.5x10^9; ETIMS 3x10^9: ETIMS: injection of peptide-coupled peripheral blood mononuclear cell (PBMC) by i.v. infusion
Period: Overall Study
Arm/Group | ETIMS 1x10^3 | ETIMS 1x10^5 | ETIMS 1x10^7 | ETIMS 1x10^8 | ETIMS 5x10^8 | ETIMS 1x10^9 | ETIMS 2.5x10^9 | ETIMS 3x10^9
Started | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ETIMS Dose Escalation: ETIMS: injection of peptide-coupled PBMC by i.v. infusion
Arm/Group | ETIMS Dose Escalation
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 42 [27 to 49]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 1
Region of Enrollment [Number; unit: participants]
  Germany | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Time Frame: 12 months
Reporting Status: Not Posted

2. Primary Outcome: Number of Adverse Events
Time Frame: 3 months after treatment
Measure: Number; unit: Number of AE
Arm/Group | ETIMS Dose Escalation
Number analyzed (Participants) | 9
Number of AE | 14

ADVERSE EVENTS:
Arm/Group | ETIMS 1x10^3 | ETIMS 1x10^5 | ETIMS 1x10^7 | ETIMS 1x10^8 | ETIMS 5x10^8 | ETIMS 1x10^9 | ETIMS 2.5x10^9 | ETIMS 3x10^9
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/2 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 1/1 | 2/2 | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETIMS 1x10^3 (N=1) | ETIMS 1x10^5 (N=1) | ETIMS 1x10^7 (N=1) | ETIMS 1x10^8 (N=1) | ETIMS 5x10^8 (N=1) | ETIMS 1x10^9 (N=2) | ETIMS 2.5x10^9 (N=1) | ETIMS 3x10^9 (N=1)
diverticulitis of sigma (Gastrointestinal disorders) | 1 (1) |  |  |  |  |  |  |
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETIMS 1x10^3 (N=1) | ETIMS 1x10^5 (N=1) | ETIMS 1x10^7 (N=1) | ETIMS 1x10^8 (N=1) | ETIMS 5x10^8 (N=1) | ETIMS 1x10^9 (N=2) | ETIMS 2.5x10^9 (N=1) | ETIMS 3x10^9 (N=1)
metallic flavor during infusion of study drug (General disorders) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Common cold (Infections and infestations) | 0 (0) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritation of punctured vein (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Vision disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0 | 0
Dysaesthesia/pain in one hand (Nervous system disorders) | 0 (0) | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric pain (Gastrointestinal disorders) | 0 (0) | 0 | 0 (0) | 0 | 1 (1) | 0 | 0 | 0
Syncope (Cardiac disorders) | 0 (0) | 0 | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0)
Paravertebral dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No